CLINICAL TRIAL: NCT01595815
Title: Successful Pregnancy and Delivery After AOA in Couples With Repeated Complete Fertilization Failure or Low Fertilization Rates
Brief Title: Successful Pregnancy and Delivery After AOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Fertility Hospital (Other)
Responsible Party: Principal Investigator, Jun-Woo Kim, Principal Investigator, Maria Fertility Hospital, Maria Fertility Hospital
Allocation: Non-Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: GJHS120509DK
Record Dates: First submitted 2012-05-09; First posted 2012-05-10 (Estimated); Last update posted 2025-05-09 (Actual); Status verified 2014-01

CONDITIONS: Infertility
Keywords: Fertilization failure, calcium ionophore, SrCl2
MeSH Terms: conditions — Infertility | interventions — Calcium Ionophores; strontium chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional ICSI (Active Comparator): The couple showed complete fertilization failure after ICSI.
  Interventions: Other: Calcium ionophore; Other: Strontium chloride (SrCl2)
- Convention ICSI (Active Comparator): The couple showed a low fertilization rates after ICSI.
  Interventions: Other: Calcium ionophore; Other: Strontium chloride (SrCl2)

INTERVENTIONS:
Other: Calcium ionophore — Oocytes were activated with calcium ionophore after ICSI
Other: Strontium chloride (SrCl2) — Oocytes were activated with strontium chloride after ICSI

SUMMARY:
Artificial oocyte activation with strontium chloride or calcium ionophore improves fertilization, embryo quality, pregnancy and delivery rate in women who showed complete fertilization failure or low fertilization rates

ELIGIBILITY:
Inclusion Criteria:

* Fertilization rate was less than 30% after conventional ICSI.
* Fertilization rate was less than 50% after ICSI with calcium ionophore.
* Repeated complete fertilization failure or low fertilization rates following ICSI in previous cycles

Exclusion Criteria:

* Fertilization rate was more than 30% after conventional ICSI
* Fertilization rate was more than 50% after ICSI with calcium ionophore.
* Successful pregnancy and delivery after ICSI in previous cycles

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2007-05; Primary Completion 2011-09 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Fertilization rate | 18 hours

SECONDARY OUTCOMES:
Embryo quality | 3 Days
Pregnancy and Implantation rates | 2 months
Assessment of Infant health care | birth and at 3, 6, 12, 24, 36, 60, and 72 months
  This assessment is according to the standard set by the National Health Insurance Service (NHIS) in Korea.

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Fertility Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim JW, Yang SH, Yoon SH, Kim SD, Jung JH, Lim JH. Successful pregnancy and delivery after ICSI with artificial oocyte activation by calcium ionophore in in-vitro matured oocytes: a case report. Reprod Biomed Online. 2015 Apr;30(4):373-7. doi: 10.1016/j.rbmo.2014.11.014. Epub 2014 Dec 11. PMID 25592974